CLINICAL TRIAL: NCT07399613
Title: Effects of Protective Step Training on Proactive and Reactive Motor Adaptations in Parkinson's Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: U.S. National Science Foundation (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00015237
Record Dates: First submitted 2024-12-12; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease; Fall; Protective Step Training; Falls, Intervention; Fall Prevention Training; Accidental Falls
Keywords: Parkinson Disease, Falls, intervention, training, Protective Step Training, accidental falls
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Crossover design:
  Prior to testing, subjects were randomly assigned to two groups. One group started with postural perturbation (PP) training (during stance), while the other group began with gait perturbation (GP) training before crossing over (during walking). During this onboarding period, self-reported and observed leg dominance in bilateral mobilizing was utilized to determine the dominant leg that will be perturbed in the walking trials. Investigators described a scenario for the participant in which they were asked which leg they would use to kick a ball over the ground.
Who Masked: Participant, Investigator
Masking Description: Randomized the all walking/training trials
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standing Perturbation Protocol (Experimental): Different postural perturbations were administered - while walking and while standing.
  Interventions: Behavioral: Protective Step Training
- Walking Perturbation Protocol (Experimental): Different postural perturbations were administered - while walking and while standing.
  Interventions: Behavioral: Protective Step Training

INTERVENTIONS:
Behavioral: Protective Step Training — Perturbation during standing and walking to actively assess proactive as well as reactive motor adaptations.
  Other Names: perturbation training; reactive step training

SUMMARY:
The aim of this study was to investigate to what extent PD affects the ability to walk, respond to balance perturbations (i.e., Protective Step Training) and produce acute short-term effects to improve compensatory reactions and control of unperturbed walking balance.

DETAILED DESCRIPTION:
Understanding the mechanism of compensation and neuroplasticity to unexpected step perturbation training during walking and static stance can have positive implications on the treatment of PD by helping to design effective training paradigms that remediate fall risk. Current rehabilitation therapies are inadequate at reducing falls in people with Parkinson's disease (PD). While pharmacologic and surgical treatments have proved largely ineffective in treating postural instability and gait dysfunction in people with PD, studies have demonstrated that therapy specifically focusing on posture, gait, and balance may significantly improve these factors and reduce falls. The primary goal of this study was to assess the effectiveness of a novel and promising intervention therapy (protective step training - i.e., PST - balance disturbance/perturbation during treadmill walking) to improve balance as measured by the reaction time and reduce falls in people with PD. A secondary goal was to understand the effects of PST on proactive and reactive feedback responses during stance and gait tasks. Multi-baseline, repeated measures analyses were performed on the multitude of proactive and reactive performance measures to assess the effects of PST on gait and postural stability parameters.

ELIGIBILITY:
Inclusion Criteria:

* able to ambulate without assistance
* had no known neurologic, cardiovascular, or orthopedic deficit - (Mini-Mental Status Examination <25), and had a Hoehn & Yahr (H&Y) score between II-III.

Exclusion Criteria:

* exhibited functionally disabling dyskinesia
* has dystonia, orthostatic hypotension,
* had neurosurgical intervention (deep brain stimulation)
* has and any significant musculoskeletal or metabolic disorders.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-03-18 (Actual)

PRIMARY OUTCOMES:
Joint (knee) reaction time | one year
  Joint (knee) Reaction time during standing and walking perturbations.

CONTACTS AND LOCATIONS:
Locations (1):
- Glencroft Senior Living: Retirement Community in Arizona, Glendale, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lockhart T, Frames C, Olson M, Moon SH, Peterson D, Lieberman A. Effects of protective step training on proactive and reactive motor adaptations in Parkinson's disease patients. Front Neurol. 2023 Oct 24;14:1211441. doi: 10.3389/fneur.2023.1211441. eCollection 2023. PMID 37965161
- See also: Frontiers Journal Manuscript — https://www.frontiersin.org/journals/neurology/articles/10.3389/fneur.2023.1211441/full